CLINICAL TRIAL: NCT07194824
Title: Design, Implementation and Analysis of a Penicillin Allergy Delabeling Model in Hospitalized Patients
Brief Title: A Penicillin Allergy Delabeling Inhospital Model Hospitalized Patients
Acronym: Des-Al-Pen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to clear evidence of the intervention's effectiveness on a pre-planned interim analysis
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/028
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Allergy Drug; Allergy Penicillin
Keywords: De-labelling; Allergy manegement; beta-lactans allergy
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Clinical evaluation study of a new care process, prospective, open, carried out in a single centre, ALTHAIA University Assistance Network of Manresa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with an active allergy label for beta-lactams admitted to hospital (Experimental): Clinical evaluation involving a review of the patient's history and a structured questionnaire, allows stratification of allergy risk into 3 categories, and managed accordingly. 1) Tipus A) Patients with a non-immune-mediated adverse reaction or with posterior tolerance. 2) Grup B) Patients with low risk potentiallly immune-mediated mechanism are considered candidates for exposure and re-exposure to penicillin and/or cephalosporins, as clinically indicted.
  3) Grup C) Patients with a previous adverse reaction considered high-risk Type C, IgE-mediated or non-immediate Type II-IV reactions,
  Interventions: Other: Pragmatic allergy management according to risk stratification

INTERVENTIONS:
Other: Pragmatic allergy management according to risk stratification — Intervention based on allergy risk stratification. Tipus A) Patients in this group can undergo direct delabeling without the need for exposure, with this being documented in the EMR. If the patient refuses, an exposure to penicillin and/or cephalosporin will be performed. Once completed, de-labeling can proceed without the need for re-exposure.
  Tipus B) Indication for use of a penicillin: Oral exposure to 250 mg of amoxicillin.
  - Indication for cephalosporin : administration of a cephalosporin that exhibits the lowest level of cross-reactivity with penicillin.
  Re-exposure to penicillin/ cephalosporin or both is performed at least 2 weeks after the first tolerated exposure. De-labeling is performed when tolerance to re-exposure is verified.
  Tipus C) These high-risk patients are managed following the protocol for the treatment of patients with beta-lactam allergy, referring them to allergy consultation for further specific test.

SUMMARY:
Design, implementation and analysis of an allergy assessment and management model beta-lactams in hospitalized patients

DETAILED DESCRIPTION:
To evaluate the impact of a healthcare process for risk stratification based on the clinical history and the application of a structured questionnaire, on the Proportion of hospitalized patients in whom the penicillin allergy label is removed

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Ability to understand the study after reading the patient information sheet (Appendix II) and providing signed consent for participation (Appendix III: informed consent form).
* Patients with a reported allergy to penicillin and/or cephalosporins that has not been investigated or with inconclusive prior testing.

Exclusion Criteria

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients hospitalized in which the penicillin allergy label is removed | At enrollment time
  Proportion of patients hospitalized in which the penicillin allergy label is removed

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Althaia, Manresa, Barcelona
  - C/ dr.Joan Soler 1-3, Manresa, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penicillin Allergy in Antibiotic Resistance Workgroup. Penicillin Allergy Testing Should Be Performed Routinely in Patients with Self-Reported Penicillin Allergy. J Allergy Clin Immunol Pract. 2017 Mar-Apr;5(2):333-334. doi: 10.1016/j.jaip.2016.12.010. No abstract available. PMID 28283158
- [Background] MacLaughlin EJ, Saseen JJ, Malone DC. Costs of beta-lactam allergies: selection and costs of antibiotics for patients with a reported beta-lactam allergy. Arch Fam Med. 2000 Aug;9(8):722-6. doi: 10.1001/archfami.9.8.722. PMID 10927711
- [Background] Macy E, Contreras R. Health care use and serious infection prevalence associated with penicillin "allergy" in hospitalized patients: A cohort study. J Allergy Clin Immunol. 2014 Mar;133(3):790-6. doi: 10.1016/j.jaci.2013.09.021. Epub 2013 Nov 1. PMID 24188976
- [Background] Gray MP, Kellum JA, Kirisci L, Boyce RD, Kane-Gill SL. Long-Term Outcomes Associated With beta-Lactam Allergies. JAMA Netw Open. 2024 May 1;7(5):e2412313. doi: 10.1001/jamanetworkopen.2024.12313. PMID 38758551
- [Background] Castells M, Khan DA, Phillips EJ. Penicillin Allergy. N Engl J Med. 2019 Dec 12;381(24):2338-2351. doi: 10.1056/NEJMra1807761. No abstract available. PMID 31826341
- [Background] Blumenthal KG, Saff RR, Banerji A. Evaluation and management of a patient with multiple drug allergies. Allergy Asthma Proc. 2014 May-Jun;35(3):197-203. doi: 10.2500/aap.2014.35.3739. PMID 24801461
- [Background] Romano A, Atanaskovic-Markovic M, Barbaud A, Bircher AJ, Brockow K, Caubet JC, Celik G, Cernadas J, Chiriac AM, Demoly P, Garvey LH, Mayorga C, Nakonechna A, Whitaker P, Torres MJ. Towards a more precise diagnosis of hypersensitivity to beta-lactams - an EAACI position paper. Allergy. 2020 Jun;75(6):1300-1315. doi: 10.1111/all.14122. PMID 31749148
- [Background] Inglis JM, Caughey GE, Smith W, Shakib S. Documentation of penicillin adverse drug reactions in electronic health records: inconsistent use of allergy and intolerance labels. Intern Med J. 2017 Nov;47(11):1292-1297. doi: 10.1111/imj.13558. PMID 28742226
- [Background] Chaudhry SB, Veve MP, Wagner JL. Cephalosporins: A Focus on Side Chains and beta-Lactam Cross-Reactivity. Pharmacy (Basel). 2019 Jul 29;7(3):103. doi: 10.3390/pharmacy7030103. PMID 31362351
- [Background] Dona I, Torres MJ, Celik G, Phillips E, Tanno LK, Castells M. Changing patterns in the epidemiology of drug allergy. Allergy. 2024 Mar;79(3):613-628. doi: 10.1111/all.15970. Epub 2023 Dec 12. PMID 38084822
- [Background] Stone CA Jr, Trubiano J, Coleman DT, Rukasin CRF, Phillips EJ. The challenge of de-labeling penicillin allergy. Allergy. 2020 Feb;75(2):273-288. doi: 10.1111/all.13848. Epub 2019 May 26. PMID 31049971
- [Background] Pano-Pardo JR, Rodilla EM, Sacristan SC, Saldana JLC, Parraga LP, Leon JLDP, Genti PR, Oviedo AR, Jaen MJT, Vidal-Cortes P, Sanz CC. Management of patients with suspected or confirmed antibiotic allergy. Executive summary of guidance from the Spanish Society of Infectious Diseases and Clinical Microbiology (SEIMC), the Spanish Society of Allergy and Clinical Immunology (SEAIC), the Spanish Society of Hospital Pharmacy (SEFH) and the Spanish Society of Intensive Medicine and Coronary Care Units (SEMICYUC). Enferm Infecc Microbiol Clin (Engl Ed). 2023 Mar;41(3):181-186. doi: 10.1016/j.eimce.2022.08.010. Epub 2023 Jan 25. PMID 36707291
- [Background] Blumenthal KG, Peter JG, Trubiano JA, Phillips EJ. Antibiotic allergy. Lancet. 2019 Jan 12;393(10167):183-198. doi: 10.1016/S0140-6736(18)32218-9. Epub 2018 Dec 14. PMID 30558872